CLINICAL TRIAL: NCT07347782
Title: Clinical Study on the Efficacy and Reliability of Speech Intelligibility Assessment for Post-stroke Patients Using an AI Solution
Brief Title: AI-Based Speech Intelligibility Assessment: Efficacy & Reliability
Acronym: AI Solution
Status: Not yet recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Prof., Pusan National University Yangsan Hospital
Other Study IDs: 11-2025-086
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Patients With Speech Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study(Patients with speech disorders)

SUMMARY:
compare the auditory-perceptual assessment conducted by speech-language pathologists using the U-TAP with the assessment performed via the AI solution (Blings) program in patients with speech disorders, and to evaluate the efficacy and reliability of these two methods for speech intelligibility assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients with neurologic disorders, including amyotrophic lateral sclerosis, poliomyelitis, cerebellar disorders, cerebellar lesions, and stroke.
* Patients presenting with concomitant speech disorders, such as dysarthria, motor speech disorders, and voice disorders.

Exclusion Criteria:

* Subjects with a score of less than 16 points on the Korean Mini-Mental State Examination (K-MMSE).
* Subjects with visual, perceptual, or auditory impairments that prevent them from following the examiner's instructions.
* Subjects judged by the researcher as unsuitable for participation in this clinical study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older with neurologic disorders-including amyotrophic lateral sclerosis (ALS), poliomyelitis, cerebellar-related disorders (such as cerebellar atrophy or degeneration and cerebellar lesions), and stroke-who present with concomitant speech disorders, such as dysarthria, motor speech disorders, and voice disorders.
  Participants must have sufficient cognitive function, defined as a Korean Mini-Mental State Examination (K-MMSE) score of 16 or higher, and must be capable of understanding and following the examiner's instructions. Individuals with visual, perceptual, or auditory impairments that interfere with participation in speech assessment, as well as those deemed unsuitable for study participation by the investigator for other clinical or practical reasons, are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Word-level consonant accuracy (%) derived from speech samples obtained during the U-TAP assessment | Visit 1 (Baseline)
  The agreement between consonant accuracy analyzed by the AI-based speech disorder analysis program (Blings) and the evaluations conducted independently by two certified speech-language pathologists (Rater 1 and Rater 2). Consonant accuracy is calculated at the word level and expressed as a percentage score ranging from 0% to 100%. The mean value of consonant accuracy scores from Rater 1 and Rater 2 is used as the reference human evaluation.

SECONDARY OUTCOMES:
Test-retest reliability of word-level consonant accuracy (%) calculated by Blings | Visit 1 and Visit 2 (7 ± 5 days interval)
  The consistency of consonant accuracy scores generated by Blings from the same participant across two visits. Comparison of Blings-derived consonant accuracy scores (%) between Visit 1 and Visit 2. Scores range from 0% to 100%.
Inter-rater agreement of word-level consonant accuracy (%) among Blings, Rater 1, and Rater 2 | Visit 1 and Visit 2 (7 ± 5 days interval)
  Agreement in consonant accuracy evaluations between the AI-based analysis and human raters. Pairwise comparisons: Rater 1 vs. Rater 2, Blings vs. Rater 1, Blings vs. Rater 2. Scores expressed as percentages (0-100%)
Time required to complete speech analysis (seconds) | Visit 1 and Visit 2 (7 ± 5 days interval)
  Comparison of analysis time between the AI-based system (Blings) and human raters. Total analysis time measured in seconds for: Rater 1, Rater 2, Blings

IPD SHARING:
Plan to Share IPD: Undecided